CLINICAL TRIAL: NCT06726616
Title: PASOS: Physical and Cognitive Aging Study in Older Adults
Brief Title: Physical and Cognitive Aging Study in Older Adults
Acronym: PASOS
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202400815
Record Dates: First submitted 2024-12-02; First posted 2024-12-10 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Older Adults (65 Years and Older); Hispanic Americans; Cognitive Aging; Aging, Healthy; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult Cohort; n=100 (50 Hispanic American adults and 50 non-Hispanic American adults): The participants in this PASOS pilot will include 50 self-identified HA individuals and 50 self-identified non-HA individuals between the ages of 55-85 years, with no psychometric evidence of neuropsychological decline. We plan to enroll an equal number of women and men. Race and ethnicity in this study will be determined via self-report or self-identification by participants.

SUMMARY:
Hispanic Americans are the fastest growing older adult group in the United States, disproportionally increasing the risk of an Alzheimer's disease and related dementias diagnosis. Efforts to reduce this risk and mitigate the related cognitive/physical declines are critical. The aim of this study is to assess the feasibility of enrolling older adults into an aging trajectory cohort, while generating preliminary data on associations of physical and cognitive aging trajectories. Our secondary objective is to generate preliminary data on the association of standard measures of physical activity and physical function with cognitive status. This study fits within our longitudinal research goal to reduce dementia incidence by understanding the mechanisms that drive the cognitive-physical aging trajectory.

DETAILED DESCRIPTION:
Overview: This study aims to assess the feasibility of recruiting and retaining 50 Hispanic American (HA) and 50 non-Hispanic American (non-HA) adults, aged 55-85, into a longitudinal aging cohort. We will evaluate differences in physical activity, physical function, and cognitive performance over time.

Design and Outcomes: Adults will be consented at the beginning of visit 1. Those potentially eligible will complete MoCA, questions about previous and current medical history, and general cognitive function (visit 1). Eligibility will be confirmed at the end of visit 1. Physical fitness, and physical activity behaviors will be assessed during visit 2. Once both visits are completed, the study team will ask about attendance availability in the future. The study team will reach out following one year (or up to 3 months after the one-year mark). The participants will be asked to repeat the same procedures as visits 1 and 2 (1 year follow-up = visits 3 and 4).

ELIGIBILITY:
Inclusion Criteria:

• Hispanic and non-Hispanic adults age 55-85 years, at least 8th grade education, community dwelling.

Additional Inclusion for Hispanic Americans

* Self-identify as Hispanic American
* Report Spanish as primary language • No evidence of dementia or mild cognitive impairment based on cognitive screening [i.e., Montreal Cognitive Assessment (MoCA) administered during Visit 1; ≥26 among non-Hispanic White, ≥25 among Hispanics, ≥24 among non-Hispanic Blacks (Milani et al., 2018)]

Exclusion Criteria:

* Inability to provide informed consent
* Artificial joint or severe disability that would make it impossible or contraindicated performing the isokinetic test
* Sensory loss (vision, hearing) or motor deficits that would preclude participation in the experimental tasks or neuropsychological assessment
* Previous major strokes or other known significant brain abnormalities or diseases affecting the brain and/or cognition (e.g., Parkinson disease, multiple sclerosis, seizure disorder, brain surgery, moderate TBI, REM Behavior Sleep Disorder, untreated sleep apnea, etc.)
* Unstable and uncontrolled medical conditions (metastatic cancer, HIV, moderate-severe kidney disease, uncontrolled diabetes, uncontrolled hypertension, severe cardiac disease, etc.). No current cancer diagnosis.
* Current or past history of major psychiatric disturbance including schizophrenia, or active psychosis, bipolar disorder, current major depressive episode, current alcohol or substance abuse or history thereof within the past six months
* Use of antipsychotics, sedatives, or other medications with significant anticholinergic properties (due to potential influence on memory)
* Use of prescribed 'memory enhancing' medications, such as Aricept or Namenda
* Previous participation in a cognitive or physical activity training study within the last 6 months or current involvement in another study involving cognitive, physical or other intervention at the time of enrollment

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hispanic Americans and Non-Hispanic American adults between the ages of 55 and 85 years old, with at least 8th grade education, and community dwelling.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2027-09-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment | From recruitment to follow-up (1-year)
  Recruiting > 80% participants (50 Hispanic American and 50 non-Hispanic American adults) for a longitudinal aging study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, College of Medicine-Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No